CLINICAL TRIAL: NCT07093333
Title: A Phase 2a, Open-label Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of ART5803 in Participants With Anti-NMDAR Encephalitis and Anti-NMDAR Antibody-Associated Psychiatric Disease
Brief Title: A Study in Participants With Anti-NMDAR Encephalitis and Anti-NMDAR Antibody-Associated Psychiatric Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arialys Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART5803-201
Record Dates: First submitted 2025-06-19; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Anti-N-methyl-D-aspartate Receptor (NMDAR) Encephalitis (ANRE); Anti-N-methyl-D-aspartate Receptor (NMDAR) Antibody-associated Psychiatric Disease; Autoimmune Encephalitis
Keywords: Anti-N-methyl-D-aspartate receptor (NMDAR); Encephalitis; Anti-N-methyl-D-aspartate receptor (NMDAR) Encephalitis
MeSH Terms: conditions — Encephalitis; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: Adult patients with chronic ANRE (Experimental)
  Interventions: Drug: ART5803
- Cohort B: Adult patients with subacute ANRE (Experimental)
  Interventions: Drug: ART5803
- Cohort C: Adult patients with acute ANRE (Experimental)
  Interventions: Drug: ART5803
- Cohort D: Adult patients with anti-NMDAR antibody-associated psychiatric disease (Experimental)
  Interventions: Drug: ART5803

INTERVENTIONS:
Drug: ART5803 — A monovalent (one-armed) antibody, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor.

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of ART5803 in adult participants with a confirmed diagnosis of anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis (ANRE) or anti-NMDAR antibody-associated psychiatric disease

DETAILED DESCRIPTION:
Anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis is one of the most common causes of autoimmune encephalitis. The disease is caused by the development of autoantibodies against the amino (N)-terminal domain (NTD) of the NMDAR subunit 1 (NR1) that bind and cross link the receptors, leading to receptor internalization and loss of function.

Arialys has developed a monovalent (one-armed) antibody, ART5803, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor. There is also an increasing body of data supporting the potential link between broader psychiatric diseases and the presence of autoantibodies against the NMDAR.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A

  1. The participant is a male or female, 18 to 65 years of age, inclusive, at the time of consent.

  2. The participant, or their legally authorized representative (LAR), must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures. For participants who are unable to sign the consent form themselves, informed consent must be obtained from their LAR in accordance with local regulations and ethical guidelines.

  3. The participant, or their LAR, must ensure willingness and ability to comply with all study procedures to the extent possible, as determined by the Investigator.

  4. The participant has a diagnosis of ANRE according to the Graus et al criteria (Graus et al, 2016), with symptom onset >9 months to ≤36 months (or ≤60 months with Sponsor approval) prior to Day 0.

  5. The participant has a positive cell-based assay result for CSF anti-NMDAR IgG antibody within 6 months of Day 0.

  6. Participants treated with IVIG must have completed treatment at least 7 days prior to Day 0.

  7. Participant receiving rituximab must be on a stable dose for at least 1 month prior to Day 0.

  8. Participants who are taking psychiatric medications (anti-depressants and anti-psychotics) must remain on stable background psychiatric medications for 4 weeks prior to Day 0 and for the first 6 weeks after Day 0.

  9. Adequate disease burden as defined as any one of the following (a to c) at Screening and Day 0:
  1. Two of the following: i. Wechsler Adult Intelligence Scale-4th Edition (WAIS-IV) immediate recall score <7 ii. Trail Making Test (TMT) Part A (TMT-A) >40 seconds iii. Rey Auditory Verbal Learning Test (RAVLT) score <7
  2. Beck Depression Inventory-II (BDI-II) total score ≥20.
  3. European Quality of Life (EuroQoL) 5 dimension, 5-level (EQ-5D-5L) score "moderate" or higher on at least 3 of the 5 items.

     10. No teratoma or removal of a teratoma at least 1 week before Screening and Day 0.

     11. Sexually active female participants of childbearing potential and male participants with female partner(s) of childbearing potential must be willing to use a highly effective method of contraception during the study (from the time of providing consent) until at least 90 days after the last study drug administration. Examples of highly effective methods of contraception are provided in Appendix 1. The contraceptive methods used for male and female participants must be documented in the source documents.

     12. Female participants of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who are surgically sterile (surgical bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) confirmed by medical history or are post-menopausal (i.e., no menstrual bleeding for more than 2 years without an alternative medical cause and confirmation with more than 1 follicle stimulating hormone [FSH] measurement of at least >40 IU/L [or higher per local institutional guidelines]).Women of non-childbearing potential are not required to use any contraceptive method.

     13. Male participants must agree not to donate sperm, and female participants must agree not to donate eggs, from the first study drug administration and until at least 90 days after the last dose of the study drug.

Cohort B and Cohort C

1. The participant is a male or female, 18 to 65 years of age, inclusive, at the time of consent.
2. The participant, or their LAR, must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures. For participants who are unable to sign the consent form themselves, informed consent must be obtained from their LAR in accordance with local regulations and ethical guidelines.
3. The participant, or their LAR, must ensure willingness and ability to comply with all study procedures to the extent possible, as determined by the Investigator.
4. The participant has a diagnosis of ANRE according to the Graus et al criteria (Graus et al, 2016), with symptom onset ≥4 months and ≤9 months (Cohort B) or ≥0 months and <4 months (Cohort C) prior to Day 0.
5. Participants with ANRE symptoms as assessed by the mRS with a score of ≥3 during Screening and Day 0.
6. The participant has a positive cell-based assay result for CSF anti-NMDAR IgG antibody within 6 months for Cohort B and 4 months for Cohort C prior to Day 0.
7. Participants treated with IVIG must have completed treatment at least 7 days prior to Day 0.
8. Participant receiving rituximab must be on a stable dose for at least 1 month prior to Day 0.
9. Participants treated with plasmapheresis must have completed treatment at least 1 day prior to Day 0.
10. Participant receiving steroids must be on a stable dose or a predefined taper regimen for at least 2 weeks prior to Day 0.
11. Sexually active female participants of childbearing potential and male participants with female partner(s) of childbearing potential must be willing to use a highly effective method of contraception during the study (from the time of providing consent) until at least 90 days after the last study drug administration. Examples of highly effective methods of contraception are provided in Appendix 1. The contraceptive methods used for male and female participants must be documented in the source documents.
12. Female participants of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who are surgically sterile (surgical bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) confirmed by medical history or are post-menopausal (i.e., no menstrual bleeding for more than 2 years without an alternative medical cause and confirmation with more than 1 FSH measurement of at least >40 IU/L [or higher per local institutional guidelines]).Women of non-childbearing potential are not required to use any contraceptive method
13. Male participants must agree not to donate sperm and female participants must agree not to donate eggs, from the first study drug administration and until at least 90 days after the last dose of the study drug.

Cohort D

1. The participant is a male or female, 18 to 65 years of age, inclusive, at the time of consent.
2. The participant, or their LAR, must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures. For participants who are unable to sign the consent form themselves, informed consent must be obtained from their LAR in accordance with local regulations and ethical guidelines.
3. The participant, or their LAR, must ensure willingness and ability to comply with all study procedures to the extent possible, as determined by the Investigator.
4. The participant has persistent psychotic symptoms for at least 2 months prior to Screening and Day 0 as evaluated by the Investigator.
5. The participant has marked deterioration of functioning in one or more areas, such as occupational, social, or personal care or hygiene.
6. The participant has the presence of:

   1. NMDAR antibodies in CSF within 6 months of Day 0 or
   2. Positive presence of anti-NMDAR antibodies in serum during Screening plus response to immune therapy or
   3. Positive CSF antibody within 12 months of Day 0 and positive serum antibody during Screening.
7. Participants treated with IVIG must have completed treatment at least 7 days prior to Day 0.
8. Participants who are taking psychiatric medications (anti-depressants and anti-psychotics) must remain on stable background psychiatric medications for at least 4 weeks prior to Day 0 and for at least the first 6 weeks after Day 0.

Adequate disease burden as defined as both of the following:

1. Subject must have a Positive and Negative Syndrome Scale (PANSS) total score ≥70 and a PANSS item score ≥4 (moderate) on 2 or more of the following PANSS items: delusions, conceptual disorganization, hallucinations, suspiciousness, and unusual thought content at Screening and Day 0.

   Exceptions may be granted on a case-by-case basis in consultation with the Sponsor.

   10. Sexually active female participants of childbearing potential and male participants with female partner(s) of childbearing potential must be willing to use a highly effective method of contraception during the study (from the time of providing consent) until at least 90 days after the last study drug administration. The contraceptive methods used for male and female participants must be documented in the source documents.

   11. Female participants of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who are surgically sterile (surgical bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) confirmed by medical history or are post-menopausal (i.e., no menstrual bleeding for more than 2 years without an alternative medical cause and confirmation with more than 1 FSH measurement of at least >40 IU/L [or higher per local institutional guidelines]).Women of non-childbearing potential are not required to use any contraceptive method.

   12. Male participants must agree not to donate sperm and female participants must agree not to donate eggs, from the first study drug administration and until at least 90 days after the last dose of the study drug

   Exclusion Criteria:

   - 1. The participant is pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.

   2. The participant has used an investigational product (IP) or investigational medical device within 30 days or 5 half-lives of the other IP (whichever is longer) prior to Screening or is required to use any investigational agent prior to completion of all scheduled study assessments.

   3. The participant has used an NMDAR modulator other than the study drug (e.g., ketamine, memantine, dextromethorphan, amantadine, ifenprodil, phencyclidine, acamprosate, D-cycloserine) from within 5 half-lives of the NMDAR modulator prior to Day 0.

   4. The participant has previous exposure to ART5803 or other antibody that targets NMDAR.

   5. Participant has any condition that, in the opinion of the Investigator, would interfere with the evaluation or administration of the IP, interpretation of participant safety or study results, or would make participation in the study an unacceptable risk.

   6. Participant with coexisting CNS demyelinating disorders (e.g., multiple sclerosis), known positivity to other antibodies associated with autoimmune encephalitis, or any significant history of a psychiatric or neurologic disorder other than ANRE should undergo consultation with the Arialys Medical Monitor on a case-by-case basis for eligibility determination.

   7. The participant has a confirmed positive test for hepatitis B serology (hepatitis B surface antigen and core antigen) and/or hepatitis C polymerase chain reaction at Screening.

   8. The participant has a history of cancer, apart from squamous cell carcinoma of the skin or basal cell carcinoma of the skin. Squamous cell and basal cell carcinomas should be treated with documented success of curative therapy >3 months prior to Screening.

   9. The participant has a history of teratoma in which teratoma has not been removed prior to entering the study. If the participant has had ovarian teratoma removed, the surgery must have occurred at least 1 week prior to Day 0. Participants with a history of malignant ovarian teratoma are excluded, irrespective of treatment. Participants with a history of associated tumors other than ovarian teratoma (e.g., other gonadal tumors) should undergo consultation with the Arialys Medical Monitor on a case-by-case basis for eligibility determination.

   10. The participant has any medical history of disease that has the potential to cause a rise in total bilirubin over the upper limit of normal. Note: Participants with a history of Gilbert's syndrome are excluded from participation from the study.

   11. The participant has a known history of allergy or reaction to any component of the investigational agent (ART5803), or history of anaphylaxis following any biologic therapy.

   12. The participant has a history of alcohol abuse or drug addiction, defined as the non-prescribed use of substances considered illegal or prohibited under the laws of the country where the trial is conducted, within the last year prior to Screening. The participant has a positive urine result for drugs of abuse (defined as any illicit drug use) at Screening or Day 0.

   13. The participant has undergone significant trauma or major surgery within 4 weeks of Screening, except for surgery to remove a teratoma.

   14. The participant has a history of herpes simplex encephalitis. 15. Participants with corrected QT interval by Fridericia (QTcF) >450 ms (males) or >470 ms (females), or QRS >120 ms. If a participant has a single ECG reading of QTcF >450 ms (males) or >470 ms (females), or QRS >120 ms the QTcF must be confirmed by averaging 3 ECGs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ART5803 | 11 weeks
  Incidence and severity of Treatment-Emergent Adverse Events (TEAEs)
To assess the safety and tolerability of ART5803 | 11 weeks
  Clinically significant changes in neurological examination findings
To assess the safety and tolerability of ART5803 | 26 weeks
  Vital signs - Systolic and diastolic blood pressure
To assess the safety and tolerability of ART5803 | 26 weeks
  Vital signs- Pulse rate
To assess the safety and tolerability of ART5803 | 26 weeks
  Vital signs- Body temperature
To assess the safety and tolerability of ART5803 | 26 weeks
  Vital signs- Respiratory rate
To assess the safety and tolerability of ART5803 | 26 weeks
  Clinical laboratory outcomes - Serum anti-ART5803 binding antibodies (ADA)
To assess the safety and tolerability of ART5803 | 11 weeks
  Concomitant medications
To assess the safety and tolerability of ART5803 | 11 weeks
  Change in suicidal tendency as measured by the incidence of positive responses (Yes) to Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) from baseline (Score range: 0-5 per item. Higher score indicated better symptoms)
To assess the safety and tolerability of ART5803 | 11 weeks
  Presence of anti-drug antibodies (ADAs)
To assess the safety and tolerability of ART5803 | Baseline
  Clinical laboratory outcomes - Alcohol Breath Drug Screen
To assess the safety and tolerability of ART5803 | Baseline
  Clinical laboratory outcomes - Urine Drug Screen
To assess the safety and tolerability of ART5803 | 26 weeks
  Clinical laboratory outcomes - Hematology
To assess the safety and tolerability of ART5803 | 26 weeks
  Clinical laboratory outcomes - Serum Chemistry
To assess the safety and tolerability of ART5803 | 11 weeks
  Clinical laboratory outcomes - Coagulation
To assess the safety and tolerability of ART5803 | 26 weeks
  Clinical laboratory outcomes - Pregnancy Test
To assess the safety and tolerability of ART5803 | Screening
  Clinical laboratory outcomes - Serology
To assess the safety and tolerability of ART5803 | Screening
  Clinical laboratory outcomes - Serum Follicle Stimulating Hormone
To assess the safety and tolerability of ART5803 | Screening
  Clinical laboratory outcomes - Urinalysis
To assess the safety and tolerability of ART5803 | Screening
  Clinical laboratory outcomes - Urine Follicle Stimulating Hormone
To assess the safety and tolerability of ART5803 | Screening
  Clinical laboratory outcomes - SARS-CoV-2 Screening
To assess the safety and tolerability of ART5803 | 26 weeks
  12-lead Electrocardiogram (ECG) findings - QTcF interval is abnormal (>450 ms for males, >470 ms for females)
To assess the safety and tolerability of ART5803 | 26 weeks
  12-lead Electrocardiogram (ECG) findings - QRS interval >120 ms

SECONDARY OUTCOMES:
To assess the effects of ART5803 on Patient Reported Outcomes (PROs) | 13 weeks
  Change from baseline in patient reported endpoints: Short Form Health Survey, Version 2 (SF-36-II) mental component domain score (Score range: 0-100. Higher score indicated better symptoms)
To assess the effects of ART5803 on Patient Reported Outcomes (PROs) | 13 weeks
  Change from baseline in patient reported endpoints: Trail Making Test, Part A (TMT-A) scores (Time to complete (higher = worse))
To assess the effects of ART5803 on Patient Reported Outcomes (PROs) | 13 weeks
  Change from baseline in patient reported endpoints: European Quality of Life, 5-dimension, 5-level (EQ-5D-5L) scores (Score range: -0.281 to 1. Higher score indicated better symptoms)
To assess the effects of ART5803 on Patient Reported Outcomes (PROs) | 13 weeks
  Change from baseline in patient reported endpoints: Beck Depression Inventory-II (BDI-II) scores (Score range: 0-63. Higher score indicated worse symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Digit Span (Score varies)
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Rey Auditory Verbal Learning Test (RAVLT) immediate recall 1 to 5 and delayed recall
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Rey-Osterrieth Complex Figure Test (36-point scoring) (ROCF-36) delayed recall component score (Score range: 0-36. Higher score indicated better symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Brief Social Aptitude Test (BSAT) number of errors
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Boston Naming Test score (Score range: 0-60. Higher score indicated better symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 13 weeks
  Change from baseline in neuropsychological endpoints: Verbal Fluency Test score (Score varies)
To assess the changes in neurological and behavioral outcomes following ART5803 administration | 13 weeks
  Time to improvement in Clinical Assessment Scale for Autoimmune Encephalitis (CASE) score by 4 points or 30% of baseline, or both. (Score range: 0-27. Higher score indicated worse symptoms)
To assess the changes in neurological and behavioral outcomes following ART5803 administration | 26 weeks
  Change from baseline in Clinical Assessment Scale for Autoimmune Encephalitis (CASE) outcomes (Score range: 0-27. Higher score indicated worse symptoms)
To assess the changes in neurological and behavioral outcomes following ART5803 administration | 16 weeks
  Change from baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score (Score range: 40-160. Higher score indicated better symptoms)
To assess changes in mobility and disability in basic and instrumental activities in daily living outcomes following ART5803 administration | 13 weeks
  In absence of rescue therapy:
  Proportion of participants with ≥1 point improvement in Modified Rankin Scale (mRS) from baseline to Week 11 Change from baseline in Modified Rankin Scale (mRS) score at Week 1, 3, and 7, and 11 as determined by rank analyses, integrating need for rescue therapy and time to achievement of the Modified Rankin Scale (mRS) Time to Modified Rankin Scale (mRS) improvement from baseline by ≥1 point (Speed of Recovery) Time to Modified Rankin Scale (mRS) ≤2
To assess the effects of ART5803 on neuropsychological assessments | 11 weeks
  Change from baseline in neuropsychological endpoints at Weeks 5 and 11:
  Positive and Negative Syndrome Scale (PANSS) score (Score range: 30-210. Higher score indicated worse symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 11 weeks
  Change from baseline in neuropsychological endpoints at Weeks 5 and 11:
  Scale for the Assessment of Negative Symptoms (SANS) score (Score range: 0-125. Higher score indicated worse symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 11 weeks
  Change from baseline in neuropsychological endpoints at Weeks 5 and 11: Clinical Global Impression-Severity (CGI-S) score (Score range: 1-7. Higher score indicated worse symptoms)
To assess the effects of ART5803 on neuropsychological assessments | 11 weeks
  Change from baseline in neuropsychological endpoints at Weeks 5 and 11:
  Change in neuropsychological endpoint Clinical Global Impression-Improvement (CGI-I) score (Score range: 1-7. Higher score indicated worse symptoms)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by maximum concentration (Cmax)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by last time point with measurable concentration (Clast)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by by last time point with minimum concentration (Cmin)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by time at which Cmax is observed (tmax)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by area under the curve from time 0 to the last measurable concentration (AUC0-t)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by area under the curve from time 0 extrapolated to infinity (AUC0-∞)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by the half-life (t½)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by the volume of distribution (Vd)
Serum PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by clearance (CL)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by maximum concentration (Cmax)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by last time point with measurable concentration (Clast)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by by last time point with minimum concentration (Cmin)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by time at which Cmax is observed (tmax)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by area under the curve from time 0 to the last measurable concentration (AUC0-t)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by area under the curve from time 0 extrapolated to infinity (AUC0-∞)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by the half-life (t½)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by the volume of distribution (Vd)
Cerebrospinal Fluid (CSF) PK parameters of ART5803 | 26 weeks
  To characterize and compare the PK profile of ART5803 as measured by clearance (CL)

OTHER OUTCOMES:
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Incidence and severity of Treatment-Emergent Adverse Events (TEAEs)
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Clinically significant changes in physical examination findings.
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Clinically significant changes in neurological examination findings
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Concomitant medications
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Change in suicidal tendency as measured by the incidence of positive responses (Yes) to Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) from baseline to multiple time points. (Score range: 0-5 per item. Higher score indicated better symptoms)
To assess the safety and tolerability of ART5803 during the Follow-up Period, after drug discontinuation | 26 weeks
  Presence of anti-drug antibodies (ADAs) at multiple time points
To assess the change in seizure frequency following ART5803 administration | 26 weeks
  Mean change in seizure frequency per 4-week period, measured from baseline (during Screening) through the end of the study as reported by seizure diary
To assess the changes in cognition following ART5803 administration | 16 weeks
  Change from baseline in Montreal Cognitive Assessment (MoCA) (Score range: 0-30. Higher score indicated better symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Sankalp Gokhale, MD, MBA, Study Chair — Arialys Therapeutics

IPD SHARING:
Plan to Share IPD: No